CLINICAL TRIAL: NCT04884997
Title: An Exploratory Study of PD-1 Antibody(Toripalimab) or Combining With Temozolomide for Injection in the Treatment of Advanced/Metastatic Malignant Melanoma
Brief Title: A Study of Toripalimab or Combining With Temozolomide（iv） in the Treatment of Advanced/Metastatic Malignant Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Yulong Zheng, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20210021C-R1
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Malignant Melanoma
Keywords: malignant melanoma; PD-1 antibody; temozolomide for injection; toripalimab
MeSH Terms: conditions — Melanoma | interventions — toripalimab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): toripalimab 3mg/kg, Q2w;
  Interventions: Drug: toripalimab
- Arm B (Experimental): toripalimab 3mg/kg, Q2w; Temozolomide 150mg/m2,d1-5,Q4w
  Interventions: Drug: toripalimab; Drug: Temozolomide Injection

INTERVENTIONS:
Drug: toripalimab — toripalimab 3mg/kg, Q2w;
  Other Names: triprizumab
Drug: Temozolomide Injection — Temozolomide 150mg/m2,d1-5,Q4w
  Other Names: Temoda
  Arms: Arm B

SUMMARY:
This study evaluate toripalimab or combining with temozolomide for injection in the treatment of advanced/metastatic malignant melanoma. Participants in arm A receive toripalimab, in arm B receive toripalimab plus temozolomide

ELIGIBILITY:
Inclusion Criteria:

* •Confirmed pathologic or cytologic diagnosis of advanced/metastatic malignant melanomawithout BRAF V600E mutation

  * ECOG PS 0-1;
  * Age :18 ~75 years old;
  * There were measurable lesions according to RECIST 1.1 and the lesions that had been irradiated showed definite progression after radiotherapy and the lesion was considered measurable only if it was not the only lesion
  * Proper function of the cardiovascular system, liver, kidney and bone marrow ;
  * Subject with at most one systemic therapy for advanced/metastatic malignant melanoma
  * Survival is expected to exceed 3 months
  * The subjects showing good compliance voluntarily participated in the study and signed the informed consent

Exclusion Criteria:

* •Previously treated with TMZ, PD-1, or PD-L1;

  * Complicated with other malignant tumors;
  * Subjects with central nervous system metastases and/or cancerous meningitis;(Unless the subjects are asymptomatic or have been treated , no radiographic evidence of new BMs or BMs enlargement is found at least 2 weeks after BMs treatment.If the subjects have active or new untreated asymptomatic central nervous system (CNS) metastases found on imaging during the screening phase,they must receive radiotherapy
  * Uncontrolled pleural effusion ,pericardial effusion or ascites requiring repeated drainage
  * Received major surgical treatment or significant traumatic injury within Random 28 days prior
  * Severe arterial/venous thrombosis events，Such as cerebrovascular accident (including temporary ischemic attack) ,deep vein thrombosis and pulmonary embolismwithin Random 6 months prior
  * Subjects with a history of psychotropic substance abuse and being unable to get rid of it or with mental disorders
  * Subjects with any severe and/or uncontrolled disease,including :

    1. Subjects with poor blood pressure control (systolic≥ 150 mmHg or diastolic ≤100mmHg)
    2. Subjects with myocardial ischemia or myocardial infarction or arrhythmia above grade I (including male QTC ≥450ms(male) and female QTC ≥470ms) And ≥grade 2 congestive heart failure (New York Heart Association (NYHA))
    3. Active or uncontrolled severe infection (≥CTC AE grade 2 infection)
    4. liver cirrhosis,active hepatitis*;*active hepatitis(Hepatitis B reference: HBsAg positive, and HBV DNA test value exceeds the normal valueHepatitis C reference: HCV antibody positive, and HCV virus titer detection value exceeds the upper limit of normal value
    5. HIV infected
    6. Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L)
    7. urine protein≥++,andConfirmated 24-hour urinary protein quantification>1.0 g
    8. Subjects received a preventive vaccineor attenuated vaccine within 4 weeks
    9. prior to first administration
    10. Participated in other clinical trials within 4 weeks
    11. Active autoimmune disease（Such as the following, but not limited to: autoimmune hepatitis interstitial pneumonia enteritis vasculitis, nephritis。Subjects with asthma requiring bronchodilators for medical intervention were not included） requiring systemic treatment（Such as the use of palliative drugs, corticosteroids, or immunosuppressants） occurred within 2 years prior to initial administration.Alternative therapy(Examples include thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) is not considered systemic therapy
    12. Other conditions that investigators consider the patients are not suitable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-07 (Actual); Primary Completion 2024-03-07 (Estimated); Study Completion 2024-09-07 (Estimated)

PRIMARY OUTCOMES:
ORR | 8 weeks
  objective response rate

SECONDARY OUTCOMES:
OS | 3 years
  overall survival
PFS | 1 years
  Progression free survival
DCR | 8 weeks
  Disease contral rate
1-year PFS | 1 year after treatment initiation
  progression free survival at 1 year (1year PFS) rate
6-month PFS | 6 months after treatment initiation
  progression free survival at 6 months (6-month PFS) rate
1-year OS | 1 year after treatment initiation
  overall survival at 1 year (1 year OS) rate
2-year OS | 2 year after treatment initiation
  overall survival at 2 years (2 year OS) rate

CONTACTS AND LOCATIONS:
Overall Officials: Yulong Zheng, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- Department of Medical Onocology, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No